CLINICAL TRIAL: NCT01180725
Title: Investigation of Dried Plums in the Treatment of Adults With Constipation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: California Dried Plum Board (Other)
Other Study IDs: Dried Plum
Record Dates: First submitted 2010-08-11; First posted 2010-08-12 (Estimated); Last update posted 2010-08-12 (Estimated); Status verified 2010-08

CONDITIONS: Constipation
Keywords: To investigate and compare the effects of dried plums and psyllium on the overall relief of constipation symptoms; To investigate and compare the taste of dried plums and psyllium; To investigate and compare the quality of life of dried plums and psyllium
MeSH Terms: conditions — Constipation | interventions — Psyllium

INTERVENTIONS:
Dietary Supplement: Dried Plum
Dietary Supplement: Metamucil

SUMMARY:
Background: Constipation is a common problem that affects nearly 60 million Americans. The treatment of constipation remains challenging with one half of patients dissatisfied with current therapy. There is a need for a food-based, natural, convenient and tasty alternative to the currently available OTC laxatives and fiber supplements, particularly for patients with occasional and mild constipation. Dried plums and prune juice have been traditionally used for the treatment of constipation but has not been systematically assessed in patients with well defined constipation. Also, the efficacy, palatability and tolerability of dried plums in the treatment of chronic constipation have not been examined.

Aim: To investigate and compare the effects of dried plums and psyllium on the overall relief of constipation symptoms, taste and quality of life in adults with functional constipation in a randomized crossover controlled trial.

Methods: We propose to study 40 subjects with functional constipation in a single blinded, randomized, cross-over study comparing 3 weeks of dried plums with 3 weeks of treatment with Psyllium

Data analysis: The primary outcome measure will be the global relief of constipation symptoms as rated by the subject at the end of each phase of the study. Additionally, we will assess several secondary outcome measures that will include the number of Complete Spontaneous Bowel Movements (CSBM) per week, Quality of Life , psychological profile, patient rating of taste on a VAS scale, patient rating of bloating, distension, satiety and fullness and patient rating of constipation-related symptoms.

Expected Results: We anticipate that treatment with dried plums will improve symptoms of constipation compared to the baseline. This improvement will be comparable to that achieved with psyllium (Metamucil) treatment. Additionally, dried plums will offer a natural, food based, convenient and more tasty alternative to over-the-counter laxatives and fiber supplements.

ELIGIBILITY:
Inclusion Criteria:

1. Constipation as defined by Rome III criteria (3,4). Patients must have symptoms for > 3 days/month for the past three months and report at least two of the following symptoms ≥ 25% of the time: straining, lumpy or hard stool, sensation of incomplete evacuation, sensation of anorectal obstruction/blockage, use of manual maneuvers, < 3 bowel movements/week. Also, they should have insufficient criteria for IBS, and only rarely experience loose stools without the use of laxatives
2. Adults between the ages of 18-75 years

Exclusion Criteria:

1. Patients taking drugs that are known to be constipating will be excluded or asked to discontinue medications for at least 2 weeks and reassessed. For example, we will recommend that patients taking calcium channel antagonists contact their respective primary care physicians to explore alternative medications for hypertension such as beta blockers or ACE-inhibitors. If the calcium channel antagonists can to be discontinued, patients will be re-screened at least two weeks after the medications are discontinued. If patients no longer meet inclusion criteria, they will be excluded from the study. Patients who remain constipated will be eligible for enrollment.
2. Patients with co-morbid illnesses such as severe cardiovascular disease, chronic renal failure, or those with previous gastrointestinal surgery except cholecystectomy and appendectomy.
3. Patients with neurologic diseases such as multiple sclerosis, strokes, spinal cord injuries, and those who have problems with cognizance, i.e. a mini-mental score of <15 and/or are legally blind will be excluded.
4. Patients with Hirschsprung' s disease, or active local anorectal problems such as anal fissures, bleeding hemorrhoids, etc
5. Patients with alternating constipation and diarrhea and those who fulfill the Rome-III criteria for irritable bowel syndrome.
6. Patients using fiber supplements, laxatives, PEG, Tegaserod or Lubiprostone and unwilling to discontinue these medications at least 2 weeks prior to the study.
7. Subjects with a known allergy to psyllium or plums.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States